CLINICAL TRIAL: NCT04187118
Title: Quality of Life in Lymphoma Patients and Cancer Care Pathway One Year Post-chemotherapy
Brief Title: Quality of Life in Lymphoma Patients One Year Post-chemotherapy
Acronym: QUALIPSO-L
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Force Hémato (Unknown); Hospitalidee (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0295
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Lymphoma
Keywords: Lymphoma; Quality Of Life; Cancer Care Pathway; Post-Chemotherapy
MeSH Terms: conditions — Lymphoma | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lymphoma patients: Patients being in complete response after a first therapy for malignant lymphoma.
  Interventions: Other: Quality of life

INTERVENTIONS:
Other: Quality of life — Quality of life one year post chemo-therapy

SUMMARY:
Malignant lymphomas are considered as among the most chemo-sensitive cancers. ML are cured in more than 85% of patient, the majority with complete response. After this active phase of treatment, patients are in "after cancer period". Toulouse University Hospital developed since 2006 the Ambulatory Medical Assistance for After Cancer program on lymphoma patient. Ambulatory Medical Assistance for After Cancer is very efficient for detecting physical and psychological complications which impact quality of life. The investigators identified 22% of lymphoma patients who had a reduced quality of life one year after the end of chemotherapy. The present study aims to investigate the evolution of observed complications and identify cancer care pathway which decrease the quality of life reduction risk in patients one year after lymphoma chemotherapy.

DETAILED DESCRIPTION:
Quality of life, as well anxiety, depression, social isolation, fear of cancer recurrence, post traumatic stress, will be measured in lymphoma patients, after a first line chemotherapy. Care cancer pathway will be also evaluated. Self-administered questionnaires will be performed on website (www.hospitalidee.fr) after inclusion and 12 months after.

ELIGIBILITY:
Inclusion Criteria:

* Patients being in complete response after a first therapy for lymphoma
* Malignant lymphoma (Hodgkin or non-Hodgkin) treated by anthracyclines with a minimum of 6 cycles, followed or not by autologous hematopoietic stem cell transplantation
* Patients informed of the study and not opposed to the research

Exclusion Criteria:

* Patients under legal guardian .
* Patients unavailable to formulate non-opposition to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life change: Quality of Life-C30 French version | Change from baseline quality of life at 12 month
  Health-related quality of life is evaluated by the use of Quality of Life-C30 French version

CONTACTS AND LOCATIONS:
Overall Officials: Loïc YSEBAERT, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No